CLINICAL TRIAL: NCT05872035
Title: Smartphone Enabled Hearing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apple Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 099-37012
Record Dates: First submitted 2023-04-26; First posted 2023-05-24 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Hearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Self-Fit Settings (Experimental): Amplification settings established by algorithm and further adjusted by participants per their preference
  Interventions: Device: Apple Software
- Pro-Fit Settings (Active Comparator): Amplification settings established by clinical reference and further adjusted by an audiologist per current best practice
  Interventions: Device: by Audiologist

INTERVENTIONS:
Device: Apple Software — Amplification settings established by algorithm and further adjusted by participants per their preference
  Arms: Self-Fit Settings
Device: by Audiologist — Amplification settings established by clinical reference and further adjusted by an audiologist per current best practice
  Arms: Pro-Fit Settings

SUMMARY:
Validation of non-inferiority between headphone amplification settings determined by a participant and settings established by audiologist best practices in individuals 18 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Proficient in written and spoken English, defined by self-report
* Mild- to moderate- hearing loss as measured by pure tone audiometry (PTA) reference test, or self-report of perceived hearing loss and 15-25 dB HL (by 4PTA)
* Participants have access to stable internet connection

Exclusion Criteria:

* Ear anatomy non-conducive to comfortable wear of headphone
* Active ear disease
* Cerumen impaction that cannot be removed
* Sudden loss of hearing (in the preceding 90 days), defined by self-report
* Self Report of loud environmental sound exposure (e.g., concert; construction site; fireworks) without hearing protection within 72 hours of reference PTA assessed at Clinic Visit 1
* Tinnitus that impacts one's daily life, defined by self-report
* Use of cochlear implants
* Self-reported issues with small or confined spaces such as a single-person enclosed booth, and/or claustrophobia
* Health technology, fitness, media outlet employees (or spouse of employees), or employees of CRO/sites contracted to execute this study
* User noted preference to not wear headphone consistently, or charge headphone and smartphone consistently, during field-use
* Hearing loss >60 dB HL at 0.25-3kHz and >65 dB HL at 4kHz in either ear; assessed during PTA
* Hearing loss that requires electroacoustic settings which are not acoustically stable in the participant's ear per audiologist judgement
* Current regular use of hearing aids
* Active treatment, or treatment in the past 6 months, with either a chemotherapeutic drug for cancer, or radiation therapy to the head or neck region
* Active treatment, or treatment in the past 6 months, with parenteral aminoglycoside antibiotics
* In the Investigator's opinion, unable to adhere to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IQVIA, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from multiple sites where audiological services were provided.
Pre-assignment Details: All 118 enrolled participants were randomized into the study
Period: Overall Study
Arm/Group | Self-Fit Settings | Pro-Fit Settings
Started | 59 | 59
Completed | 59 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-Fit Settings | Pro-Fit Settings | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 68
  >=65 years | 26 | 24 | 50
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at Birth
  Participants
    Female | 30 | 39 | 69
    Male | 29 | 20 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 58 | 58 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 10 | 14
  White | 53 | 48 | 101
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Geographical Region of Recruitment and Enrollment
  Participants
    United States | 59 | 59 | 118
Subject Medical History with >10.0% Occurrence [Count of Participants; unit: Participants] — Medical history affecting at least 10% of study participants in any treatment group
  Participants
    Deafness bilateral | 26 | 23 | 49
    Hypertension | 10 | 12 | 22
    Hypoacusis | 5 | 6 | 11
    Tinnitus | 14 | 4 | 18
Four-Frequency Pure Tone Average Results-Full Analysis Set [Count of Participants; unit: Participants] — Classification of the reference audiometry values averaged across four frequencies (0.5, 1, 2, and 4 kHz)
  Participants
    15-25 dB HL (No Impairment) | 12 | 15 | 27
    26-40 dB HL (Mild Impairment) | 26 | 26 | 52
    41-60 dB HL (Moderate Impairment) | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: International Outcome Inventory for Hearing Aids (IOI-HA) Survey Results
Description: The IOI-HA survey is a 7-item questionnaire that assesses the effectiveness of hearing aids. It was self-administered to each study participant one time at the third scheduled clinic visit approximately 18-31 days after enrollment. For each participant, the IOI-HA total score (which ranges from 7-35 where higher scores indicate a better outcome) was computed and the mean IOI-HA scores were compared between the Experimental and Reference Groups.
Time Frame: Approximately 18-31 days upon enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-Fit Settings | Pro-Fit Settings
Number analyzed (Participants) | 59 | 59
score on a scale | 25.5 (3.03) | 26.6 (3.63)

ADVERSE EVENTS:
Time Frame: Participants were evaluated by the PI and/or designee(s) at each of the three scheduled clinic visits from the time they signed the ICF until they completed the study (approximately 18-31 days after enrollment).
Arm/Group | Self-Fit Settings | Pro-Fit Settings
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 1/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-Fit Settings (N=59) | Pro-Fit Settings (N=59)
Chest Pain (General disorders) | 0 (0) | 1 (1) — Unspecified chest pain
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Painful left arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT05872035/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT05872035/SAP_001.pdf